CLINICAL TRIAL: NCT06691464
Title: [68Ga]-FAPI PET/CT to Detect Fibroblast Activity in Non-resolving ARDS, a Feasibility Study.
Brief Title: FAPI PET/CT to Detect Fibroblast Activity in Non-resolving ARDS
Acronym: FAPI ARDS
Status: Enrolling by invitation | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 11304; 2024-517257-27-00 (EU CTIS Number); 2022-003701-29 (EudraCT Number); Review board UMCG (Registry Identifier: 2022/577); CCMO (Registry Identifier: NL83114.042.22)
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-10

CONDITIONS: ARDS (Moderate or Severe)
Keywords: ARDS; respiratory failure; FAPI; PET/CT
MeSH Terms: conditions — Lymphoma, Follicular; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Broncho alveolair lavage (BAL) for respiratory cytology allowing for scRNA analysis.
  Blood serum and plasma. Nose swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: PET — FAPI - PET/CT

SUMMARY:
Of patients requiring mechanical ventilation in the ICU 23% meet criteria of the Acute Respiratory Distress Syndrome (ARDS). Mortality of this syndrome remains high (35-46%) in moderate and severe ARDS. In patients not recovering from ARDS, fibroblasts seem to play an important role. However, the effect of fibroblast activity on the lack of pulmonary recovery is not fully understood. The new PET tracer [68Ga]FAPI-46 (FAPI) allows for imaging of activated fibroblasts. The aim of this study is to explore the pulmonary fibroblast activity, measured with the FAPI PET/CT, in patients with non-resolving ARDS.

DETAILED DESCRIPTION:
Of patients requiring mechanical ventilation in the ICU 23% meet criteria of the Acute Respiratory Distress Syndrome (ARDS). Mortality of this syndrome is high (35-46%) in moderate and severe ARDS. The fibroproliferative phase plays an important role in patients not recovering from ARDS. Bronchoalveolar lavage (BAL) can be used to investigate this process. However, quantitative assessment using BAL of fibroblast activity in both lungs is invasive, indirect and has yielded inconsistent results. This has precluded clinical utility. New methods to assess fibroblast activity in ARDS are therefore needed. A novel tool is PET/CT with the tracer [68Ga]-FAPI-46. [68Ga]-FAPI PET has the ability for reproducible and non-invasive measurement of fibroblast activity.

Objective:

1. To relate pulmonary fibroblast activity in non-resolving ARDS, measured by FAPI-PET/CT, to 28 day mortality, ventilator-free days and alive at 28 days (VFD-28) and ICU length of stay.
2. To study the relationship between pulmonary fibroblast activity and systemic fibrotic and inflammatory biomarker.
3. To relate the pulmonary fibroblast activity on [68Ga]FAPI PET/CT with respiratory cell phenotypes and fibrotic and inflammatory mediators collected via bronchoalveolar lavage (BAL).

Study design: This is a single center prospective observational feasibility study. We will include 20 ventilated patients with non-resolving ARDS. All mechanically ventilated patients in the ICU will be screened daily for ARDS. When ARDS is present for 5 consecutive days, patients will be included. Within 7 days after inclusion a [68Ga]FAPI-46 PET/CT scan will be performed. Within 48 hours of the PET/CT a broncho alveolar lavage and a nasal brush, will be performed. Blood will be drawn at inclusion and every 3rd day, as well as the day of the PET/CT. Daily registration of ventilatory and circulatory parameters, as well as clinical blood parameters, will be collected.

End of study: The study will end when the patient has died, is discharged from the ICU or after 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated
* Patient meets the criteria for non-resolving ARDS as at day 5 of the ARDS diagnosis one or more of the following criteria is true:

  * P/F ratio <200 mmHg
  * Positive End Expiratory Pressure (PEEP) of 12 cmH2O or more
  * Static lung compliance of < 50 ml/cmH2O
* Deemed safe for transport by attending clinician (staff Intensivist)
* Informed consent signed by patient or legal representative

In case of COVID-19 a SARS-CoV-2 PCR CT of > 30 is required.

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Inability to attain informed consent
* Too unstable for transport as judged by the treating staff intensivist

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU who are mechanically ventilated and fulfil the ARDS criteria for more than 5 days.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Patient outcome - ICU stay | From inclusion until the end of the study (28 days after inclusion)
  Pulmonary FAP expression, measured by [68Ga]-FAPI PET/CT, correlated to 28 days of ICU stay.
Patient outcome - 28 days mortality | From inclusion until end of the study (28 days after inclusion)
  Pulmonary FAP expression, measured by [68Ga]-FAPI PET/CT, correlated to 28 days mortality.
Patient outcome - VFD-28 | From inclusion until end of the study (28 days after inclusion)
  Pulmonary FAP expression, measured by [68Ga]-FAPI PET/CT, correlated to ventilation free days of 28 days (VFD-28)

SECONDARY OUTCOMES:
Systemic ECM and inflammatory markers | On day of PET/CT
  Pulmonary FAP expression, measured by [68Ga]-FAPI PET/CT, correlated to extra cellular matrix and inflammatory parameters on the day of PET/CT.
Respiratory ECM and inflammatory markers | within 48 hours before or after PET/CT
  Pulmonary FAP expression, measured by [68Ga]-FAPI PET/CT, correlated to BAL extra cellular matrix, inflammatory parameters and cellular phenotypes
Respiratory scRNA | within 48 hours before or after PET/CT
  Around the time of the PET/CT a broncho alveolair lavage will be performed collecting respiratory system cells which will be analysed using scRNA analysis.

OTHER OUTCOMES:
Nasal brush scRNA | 48 hours before or after the PET/CT
  scRNA of the BAL will be correlated to the scRNA of the nasal brush.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided